CLINICAL TRIAL: NCT03159988
Title: Angiotensin (1-7) Treatment to Improve Cognitive Functioning in Heart Failure Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Suspended. Slow enrollment.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Meredith Hay, Professor, University of Arizona College of Medicine Department of Physiology and Department of Psychology; Evelyn F. McKnight Brain Institute, Sarver Heart Center University of Arizona, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510150837
Record Dates: First submitted 2016-10-23; First posted 2017-05-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — angiotensin I (1-7); Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Non-randomized treatment group (Experimental): 12 weeks of daily does subcutaneous injection of Angiotensin-(1-7) 100 mcg/kg/day
  Interventions: Drug: Angiotensin-(1-7); Behavioral: Memory Training

INTERVENTIONS:
Drug: Angiotensin-(1-7) — Angiotensin-(1-7) 100mcg/kg/day for 12 weeks
Behavioral: Memory Training — 50% of the treatment arm will receive 2 session per week for 2 weeks of memory training

SUMMARY:
Heart failure (HF) is the major cardiovascular disease that continues to grow in prevalence, largely due to aging of the population. HF is described as the inability of the heart to keep up with the demands on it and, specifically, failure of the heart to pump blood with normal efficiency. Cognitive impairment (CI) is common in HF patients, resulting in a person having trouble remembering, learning new things, concentrating, or making decisions that affect their everyday life. Patients with HF have been show repeatedly to have trouble remembering and learning new things when compared to the general population. Patients with demonstrated CI have a significantly increased risk of developing dementia (memory loss). It is believed that the reason HF patients have a higher risk of CI is possibly due to less blood reaching the brain and an overall inflammatory process occurring in the body including the brain. To date there are no known therapies that can help treat CI caused by HF.

A substance, Angiotensin-(1-7) [Ang-(1-7)], is known to decrease inflammation in the brain. Early studies in humans have shown it to be safe. This substance is naturally produced in the body and works by activating areas in the brain involved in memory. Investigators believe that Ang-(1-7) may be able to help lower the risk of loss of cognitive function in patients with heart failure.

In this study, we will try to determine whether Ang-(1-7) is a safe and effective treatment for cognitive impairment in HF patients.

DETAILED DESCRIPTION:
In this non-randomized pilot study 16 heart failure patients will be enrolled. Adults (ages 55-75) with chronic HF will be recruited who do not have neurologic or psychiatric disorders expected to interfere with memory function. Patients must have been diagnosed with HF ≥ 90 days prior to enrollment, be clinically stable, and on stable medications. Participants have a medical history and examination, with documentation of evidence of HF, and screening to rule out dementia (Mini-Mental State Exam score less than 25), and depression (Geriatric Depression Scale score greater than 10. Participants will be treated for 12 weeks with a daily dose of subcutaneous Ang-(1-7) (100 mcg/kg/day). Half of the group will be given memory training in 2-hr sessions twice weekly for two weeks beginning at 6 weeks of drug treatment. Prior to drug treatment, baseline measures will include memory and neuropsychological tests and inflammatory markers. Memory and neuropsychological tests will be repeated at 3 weeks, 6 weeks and 12 weeks. Inflammatory biomarkers will be reassessed at 6 weeks and 12 weeks. Blood draws for pharmacokinetic (PK) measurements will be obtained at baseline and Day 7. MRI scans will be obtained from all participants who do not have an ICD, pacemaker or other contraindication to MRI at baseline with repeat scans at 12 weeks. Lastly Self-Care Efficacy testing will be obtained at 12 weeks from all participants.

Aim 1 Primary Outcome: Changes in performance on the Memory Intentions Test (MIST, a test of PM) between baseline and 12 weeks27 will be the primary endpoint to test effectiveness of PMT in the presence or absence of Ang-(1-7) treatment.MIST scores have been shown to predict medication adherence.

Aim 1 Secondary Outcomes:

1. Safety of the treatment will be assessed by careful collection of standard serious adverse events, and comparison of events across treatment arms. In addition, patients will be asked about difficulties associated with the therapy, and medication vials collected to assess compliance with therapy.
2. Self-care efficacy at 12 weeks will be measured using the SCHFI, a validated tool.
3. Other neuropsychological measures of memory, executive functions, and psychomotor speed will be assessed at baseline, 3 weeks, 6 weeks, and at the 12 week follow-up.
4. HF quality of life will be assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at baseline and 12 weeks.
5. Adjudicated HF hospitalizations, all-cause hospitalizations and death will be assessed by treatment arm.

Aim 2: Systemic Inflammation Assay: At baseline, and after 6 and 12 weeks of Ang-(1-7) treatment, blood will be collected for assessment of systemic inflammation. Blood will be placed in lavender-top EDTA tubes, centrifuged to obtain plasma, and rapidly frozen in liquid nitrogen.

Cytokines, chemokines, and additional circulating inflammatory analytes will be detected and quantified by multiplex immunoassay using a MAGPIX®. Each sample will be measured in duplicate. Data will be analyzed by ANOVA across all groups.

Aim 2 Primary Outcome: Immunosuppressive cytokines TGFα and IL-1 will be measured as they play an important role in the anti-inflammatory actions of Ang-(1-7) and are widely used as functional indicators of systemic inflammation. The more common clinical inflammatory marker of systemic inflammation C-reactive protein, will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic HF ≥ 90 days prior to enrollment
* Be clinically stable and on stable medications
* Stable NYHA Class II-III HF or symptoms during mild or moderate exercise but not at rest (i.e. shortness of breath)
* Fluent in English or formal education in English starting from at least the age of 5
* Able and willing to provide informed consent

Exclusion Criteria:

* Evidence of decompensated HF
* Symptoms or signs of active coronary ischemia
* Criteria for DSM-IV diagnosis or history of serious psychiatric disease, or diagnosed learning disabilities. May have psychological problem that has been well controlled on medication for a sustained period of more than 2 years.
* Any other neurological, psychiatric, or medical illness or injury expected to interfere with cognitive function or memory including but not limited to stroke (diagnosed with evidence of stroke), head injury, epilepsy, Alzheimer's, Parkinson's, brain cancer, depression (current, but ok in past). Migraines OK. May have TIAs with no sign of impairment and no sequelae following the event
* Active substance abuse disorder i.e. alcohol, nicotine. Previous substance abuse of cocaine, Ecstasy, LSD, IV drugs
* History of seizure disorder as child or currently experiencing or on medications for seizures. Exception is febrile seizures as a child.
* Any condition which may prevent the subject from adhering to the study protocol, as determined by the Investigator i.e. reported learning disability, cataracts impairing vision, colorblindness.
* Movement disorders that prevent the subject from being still for the MRI
* The presence of any metallic implant or foreign body, including dental bridges excludes patients from MRI. Removable body piercings/implants okay. Patients with a metal implant or foreign body will still be enrolled; however these patients will not undergo MRI testing.
* Professional metalworker or welder
* Recurring panic attacks or claustrophobic
* Abnormally high weight or height to fit in scanner (Bore 70cm)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04; Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in performance on the Memory Intentions Test (MIST) | Baseline and 12 weeks
  MIST will be performed at baseline and 12 weeks to test prospective memory

SECONDARY OUTCOMES:
Assessment of self-reported Quality of Life (QoL) | Baseline and 12 weeks
  Assessment of QoL will be performed at baseline and 12 weeks utilizing the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Systemic Inflammation Assay | 6 weeks and 12 weeks
  Assessment of systemic inflammation will be performed using plasma samples at 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Sarver Heart Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided